CLINICAL TRIAL: NCT00281697
Title: A Phase III, Multicenter, Randomized, Placebo-controlled Trial Evaluating the Efficacy and Safety of Bevacizumab in Combination With Chemotherapy Regimens in Subjects With Previously Treated Metastatic Breast Cancer
Brief Title: A Study to Evaluate the Safety and Efficacy of Bevacizumab in Combination With Chemotherapy in Previously Treated Metastatic Breast Cancer (RIBBON 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVF3693g
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Results first posted 2012-09-24 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Metastatic Breast Cancer
Keywords: Ribbon 2; Avastin; MBC; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Standard chemotherapy + bevacizumab (Experimental): Patients received one of several standard chemotherapies for metastatic breast cancer plus bevacizumab in a dose of either 10 mg/kg intravenously (IV) every 2 weeks or 15 mg/kg IV every 3 weeks depending upon the schedule of chemotherapy chosen.
  Interventions: Drug: Bevacizumab; Drug: Standard chemotherapy
- Standard chemotherapy + placebo (Placebo Comparator): Patients received one of several standard chemotherapies for metastatic breast cancer plus placebo to bevacizumab administered IV either every 2 weeks or every 3 weeks depending upon the schedule of chemotherapy chosen.
  Interventions: Drug: Placebo; Drug: Standard chemotherapy

INTERVENTIONS:
Drug: Bevacizumab — The dose of bevacizumab was based on a patient's weight at baseline and remained the same throughout the study.
  Other Names: Avastin
  Arms: Standard chemotherapy + bevacizumab
Drug: Placebo
  Arms: Standard chemotherapy + placebo
Drug: Standard chemotherapy — Patients received one of the following four standard chemotherapies for metastatic breast cancer.
  1. Taxane - Paclitaxel (Taxol) 90 mg/m^2 IV every week for 3 weeks followed by 1 week of rest; paclitaxel (Taxol) 175 mg/m^2 IV every 3 weeks, or paclitaxel protein-bound particles (Abraxane) 260 mg/m^2 IV every 3 weeks; or docetaxel (Taxotere) 75-100 mg/m^2 IV every 3 weeks.
  2. Gemcitabine (Gemzar) 1250 mg/m^2 IV on Days 1 and 8 of each 3-week cycle.
  3. Vinorelbine (Navelbine) 30 mg/m^2 IV every week of each 3-week cycle.
  4. Capecitabine (Xeloda) 1000 mg/m^2 orally twice daily on Days 1-14 of each 3-week cycle.

SUMMARY:
This phase III, multicenter, randomized, placebo-controlled, blinded trial is designed to evaluate the efficacy and safety of bevacizumab when combined with standard chemotherapy compared with chemotherapy alone in subjects with previously treated metastatic breast cancer.

DETAILED DESCRIPTION:
For all Outcome Measures except Overall Survival and One-year Survival, the Time Frame was from Baseline to data cut-off for analysis of the primary Outcome Measure (up to 3 years 2 months). For the Outcome Measures Overall Survival and One-year Survival, the Time Frame was from Baseline to the end of the study (up to 6 years, 7 months).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* ≥ 18 years of age.
* Histologically confirmed carcinoma of the breast with measurable or non-measurable metastatic disease that has progressed (patients with a history of brain metastasis are eligible for study participation [USA only], as long as their brain metastases have been treated and they have no evidence of progression or hemorrhage after treatment and no ongoing requirement for dexamethasone).
* Progression of disease during or following administration of one (non-investigational) chemotherapy regimen administered in the first-line setting.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* For women of childbearing potential, use of an effective means of non-hormonal contraception.
* Life expectancy ≥ 3 months.
* Willingness and capacity to comply with study and follow-up procedures.

Exclusion Criteria:

* Prior hormonal therapy only as treatment for metastatic disease without chemotherapy. Patients must have received chemotherapy for their metastatic disease in the first-line setting. Hormone therapy alone is not allowed.
* For subjects who have received prior anthracycline-based therapy, documentation of left ventricular ejection fraction < 50% by either multiple gated acquisition (MUGA) or echocardiogram (ECHO).
* Treatment with more than one prior cytotoxic regimen for metastatic breast cancer (MBC).
* HER2-positive status (patients who have unknown HER2 status, and for whom determination of HER2 status is not possible, are eligible for this study).
* Unknown estrogen receptor (ER) and progesterone receptor (PR) status.
* Radiation therapy other than for palliation or brain metastasis, biologic therapy, or chemotherapy for MBC within 21 days prior to Day 0 (Day 1 of Cycle 1 of treatment).
* Prior therapy with bevacizumab or other vascular endothelial growth factor (VEGF) pathway-targeted therapy.
* Untreated brain metastasis.
* Inadequately controlled hypertension.
* Unstable angina.
* New York Heart Association Grade II or greater congestive heart failure (CHF).
* History of myocardial infarction within 6 months prior to Day 0 (the day of the first bevacizumab/placebo infusion).
* History of stroke or transient ischemic attack within 6 months prior to Day 0.
* Clinically significant peripheral vascular disease.
* Evidence of bleeding diathesis or coagulopathy.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0; anticipation of need for major elective surgical procedure during the study.
* Minor surgical procedures, fine-needle aspirations, or core biopsies within 7 days prior to Day 0.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0.
* Serious, non-healing wound, ulcer, or bone fracture.
* History of anaphylactic reaction to monoclonal antibody therapy not controlled with treatment premedication.
* History of other malignancies within 5 years of Day 0, except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* inadequate organ function.
* Pregnancy (positive serum pregnancy test) or lactation.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the subject at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2006-02; Primary Completion 2009-03 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo Faoro, MD, Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Chemotherapy + Bevacizumab | Standard Chemotherapy + Placebo
Started | 459 | 225
Completed | 58 | 28
Not Completed | 401 | 197
Not completed — > 60 days since last dose of study drug | 4 | 4
Not completed — Adverse Event | 54 | 15
Not completed — Death | 8 | 3
Not completed — Disease progression | 279 | 149
Not completed — Other | 5 | 6
Not completed — Physician's decision to withdraw | 15 | 12
Not completed — Subject/guardian's decision to withdraw | 33 | 6
Not completed — Did not receive study drug | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Chemotherapy + Bevacizumab | Standard Chemotherapy + Placebo | Total
Number analyzed (Participants) | 459 | 225 | 684
Age Continuous [Mean (Standard Deviation); unit: years] | 55.6 (11.0) | 55.0 (11.2) | 55.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 457 | 225 | 682
  Male | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: PFS was defined as the time from randomization to first documented disease progression (PD) as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) or death due to any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions. Target lesions should be selected on the basis of their size (those with the longest diameter) and their suitability for accurate repeated measurements by imaging techniques or clinically. All measurable lesions up to a maximum of 5 lesions per organ and 10 lesions in total, representative of all involved organs, should be identified as target lesions.
Time Frame: Baseline to data cut-off for analysis of the primary Outcome Measure (up to 3 years, 2 months)
Population: Intent-to-treat population: All randomized patients, regardless of whether they received any study drug or completed the full course of treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard Chemotherapy + Bevacizumab | Standard Chemotherapy + Placebo
Number analyzed (Participants) | 459 | 225
Months | 7.2 [6.5 to 7.6] | 5.1 [4.1 to 6.0]

2. Secondary Outcome: Progression-free Survival Within Individual Standard Chemotherapy Cohorts (Taxanes, Gemcitabine, Capecitabine, and Vinorelbine)
Description: Progression-free survival was defined as the time from randomization to first documented disease progression as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) or death due to any cause, whichever occurred first. Results are reported for each of the 4 standard chemotherapy cohorts used in the study.
Time Frame: Baseline to data cut-off for analysis of the primary Outcome Measure (up to 3 years, 2 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard Chemotherapy + Bevacizumab | Standard Chemotherapy + Placebo
Number analyzed (Participants) | 459 | 225
Months
  Taxanes, n=201, 103 | 8.0 [7.2 to 9.3] | 5.8 [4.2 to 7.9]
  Gemcitabine, n=108, 52 | 6.0 [5.5 to 7.1] | 5.5 [2.6 to 7.5]
  Capecitabine, n=97, 47 | 6.9 [5.5 to 8.5] | 4.1 [2.8 to 5.1]
  Vinorelbine, n=53, 23 | 5.7 [3.5 to 7.5] | 7.0 [2.7 to 8.9]

3. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization to death from any cause.
Time Frame: Baseline to the end of the study (up to 6 years, 7 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard Chemotherapy + Bevacizumab | Standard Chemotherapy + Placebo
Number analyzed (Participants) | 459 | 225
Months | 18.6 [17.4 to 20.0] | 17.8 [15.1 to 20.4]

4. Secondary Outcome: One-year Survival
Description: Percentage of patients who survived 1 year in the study.
Time Frame: Baseline to the end of the study (up to 6 years, 7 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Standard Chemotherapy + Bevacizumab | Standard Chemotherapy + Placebo
Number analyzed (Participants) | 459 | 225
Percentage of patients | 70.5 [66.3 to 74.7] | 68.6 [62.5 to 74.8]

5. Secondary Outcome: Objective Response
Description: A patient had an objective response if they had a complete response or a partial response determined on two consecutive occasions ≥ 4 weeks apart as determined by the investigator using RECIST. For target lesions, a complete response was defined as the disappearance of all target lesions; a partial response was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. For non-target lesions, a complete response was defined as the disappearance of all non-target lesions; a partial response was defined as the persistence of 1 or more non-target lesions.
Time Frame: Baseline to data cut-off for analysis of the primary Outcome Measure (up to 3 years, 2 months)
Population: Intent-to-treat population: All randomized patients, regardless of whether they received any study drug or completed the full course of treatment. Only patients who had measurable disease at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Standard Chemotherapy + Bevacizumab | Standard Chemotherapy + Placebo
Number analyzed (Participants) | 362 | 179
Percentage of patients | 39.5 [34.4 to 44.7] | 29.6 [23.0 to 36.7]

6. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response was defined as the time from the initial response to documented disease progression or death from any cause, whichever occurred first. Duration of objective response was only analyzed in patients who achieved an objective response.
Time Frame: Baseline to data cut-off for analysis of the primary Outcome Measure (up to 3 years, 2 months)
Population: Intent-to-treat population: All randomized patients, regardless of whether they received any study drug or completed the full course of treatment. Only patients who had measurable disease at baseline and achieved an objective response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Standard Chemotherapy + Bevacizumab | Standard Chemotherapy + Placebo
Number analyzed (Participants) | 143 | 53
Months | 7.3 [6.2 to 8.2] | 7.5 [6.6 to 9.2]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline to the end of the study (up to 6 years, 7 months).
Description: Adverse events are reported for safety-evaluable population defined as all randomized patients who received study treatment, defined as at least 1 full or partial dose of bevacizumab, placebo, or standard chemotherapy.
Arm/Group | Standard Chemotherapy + Bevacizumab | Standard Chemotherapy + Placebo
Serious Adverse Events (participants affected / at risk) | 112/458 | 39/221
Other Adverse Events (participants affected / at risk) | 125/458 | 39/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Chemotherapy + Bevacizumab (N=458) | Standard Chemotherapy + Placebo (N=221)
Vomiting (Gastrointestinal disorders) | 6 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Periproctitis (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 3
Infection (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 3
Bronchitis (Infections and infestations) | 2 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 5
Neutropenia (Blood and lymphatic system disorders) | 6 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Fascitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 2
Asthenia (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 1
Thrombosis in device (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Performance status decreased (General disorders) | 1 | 0
Sudden death (General disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Superior vena caval syndrome (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 1 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Cranial nerve paralysis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 2
Pericardial effusion (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 3 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 1
Conversion disorder (Psychiatric disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Embolism (Vascular disorders) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0
Device dislocation (General disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Chemotherapy + Bevacizumab (N=458) | Standard Chemotherapy + Placebo (N=221)
Neutropenia (Blood and lymphatic system disorders) | 77 | 33
Peripheral sensory neuropathy (Nervous system disorders) | 25 | 9
Hypertension (Vascular disorders) | 37 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.